CLINICAL TRIAL: NCT03740685
Title: Changes in High Sensitive C Reactive Protien With Different Treatment Modalities in Acute Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelhamed, principal investigator, Assiut University
Other Study IDs: CHCPWDTM
Record Dates: First submitted 2018-10-11; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Pancreatitis, Acute
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute pancreatitis: All patients will recive different lines of treatment {saline,antibiotics,dexamethasone}
  Interventions: Diagnostic Test: High sesitive C reactive protien

INTERVENTIONS:
Diagnostic Test: High sesitive C reactive protien — High sesitive C reactive protien will be evaluated at admission time and after 36 hours

SUMMARY:
changes in high sensitive C reactive protien with different treatment modalities in acute pancreatitis

ELIGIBILITY:
Inclusion Criteria:

* Age>=18 years
* Diagnosis of acute pancreatitis confirmed by at least 2 of the following:

  1. Typical epigastric abdominal pain
  2. Elevation amylase/lipase >3 times upper limit normal and/or
  3. Confirmatory findings on cross-sectional imaging
  4. Enrollment within 8 hours of presentation

Exclusion Criteria:

* Class II or greater NYHA heart failure
* Oxygen dependent COPD
* Chronic kidney disease>stage 2
* Existing necrosis on abdominal CT
* Organ dysfunction prior to enrollment
* Sepsis
* Acute respiratory distress syndrome
* Malignancy not in remission for at least 5 years
* Active drug use
* Known allergy to dexamethasone
* Altered mental status
* Insulin-requiring diabetes
* Abdominal surgery within 60days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute pancreatitis
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-11-09 (Estimated); Primary Completion 2018-11-09 (Estimated); Study Completion 2019-10-08 (Estimated)

PRIMARY OUTCOMES:
High sesitive C reactive protien | 72hours
  Level of High sesitive C reactive protien expected to be changed with different lines of treatment and will be compaered
Serum Amylase | 72hours
  Level of Serum Amylase expected to be changed with different lines of treatment and will be compaered
Serum Lipase | 72hours
  Level of Serum Lipase expected to be changed with different lines of treatment and will be compaered

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No